CLINICAL TRIAL: NCT04900506
Title: Cemented Hemiarthroplasty in Femoral Neck Fractures; Are Clinical Results Affected by Surgical Approach. A Randomized Clinical Trial Comparing Posterior and Anterior Approach
Brief Title: Surgical Approach in Hemiarthroplasty. A Randomized Clinical Trial Comparing Posterior and Anterior Approach
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Sorlandet HF
Record Dates: First submitted 2021-05-05; First posted 2021-05-25 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-11

CONDITIONS: Femoral Neck Fractures; Bone Mineral Density; Muscle Damage; Surgical Approach
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Bone Density

STUDY DESIGN:
Intervention Model Description: Patients are allocated to either an anterior approach or a posterior approach after inclusion. Both groups are operated with a cemented hemiarthroplasty
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Outcome assessors are blinded to allocation by not having access to patients study protocol and by examining patients covering their operated hip with clothing.
  Patients are attempted blinded by using wound dressings to cover their operated hip and are, unless expressing specific interest in knowing the surgical approach, not informed of the randomization result. To evaluate the blinding of patients we will record their knowledge of which surgical approach they were operated with at their 12-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cemented hemiarthroplasty , posterior SPAIRE approach (Active Comparator): Posterior SPAIRE approach: lateral decubitus position, preservation of the piriformis tendon and obturator internus, detatchment of obturator externus , capsular T-incision, femoral neck resection, femoral canal reaming according to preoperative templating, third generation cementation technique, capsular repair, repair of obturator externus.
  Interventions: Procedure: Posterior SPAIRE approach, anterior approach
- cemented hemiarthroplasty, anterior approach (Active Comparator): Anterior approach: supine position, both legs washed and draped, intermuscular plane between m. tensor fascia lata and m. sartorius, capsular T-incision, femoral neck resection, femoral canal reaming according to preoperative templating, third generation cementation technique, capsular repair
  Interventions: Procedure: Posterior SPAIRE approach, anterior approach

INTERVENTIONS:
Procedure: Posterior SPAIRE approach, anterior approach — Based on power calculation a sub-group analysis of 50 patients will be examined with DXA, all patients for biochemical and clinical muscle damage (CK, CRP, TUG-test, Trendelenburg, strenght test)
  Other Names: Bone Mineral Density; Biochemical muscle damage; Clinical muscle damage

SUMMARY:
Dislocated femoral neck fractures are routinely treated with cemented hemiartroplasty and the direct lateral approach (Hardinge) has commonly been used in Norway. The investigators have lately witnessed a significant change in the prefered surgical approaches in total hip arthroplasty (THA) in favor of the posterior and anterior approaches. The direct lateral approach has in THA, more or less, been abandoned in Norway. Numerous studies have reported superior results using the posterior and anterior approahes compared to the lateral approach.

DETAILED DESCRIPTION:
The investigators have witnessed a marked change in preferred anatomical route to the hip joint when performing total hip artrhroplasty (THA) for osteoarthritis in Norway. The direct lateral approach, which 10 years ago dominated, is today more or less abandoned. Several studies have reported inferior results in patients operated with the lateral approach compared to the posterior and anterior approaches, the latter approaches used in approximately 95 % of all THA´s i Norway. Many approaches are known for hip arthroplasty in trauma patients, but there is little consensus on the preferred method. The preferred surgical approach varies among hospitals and surgeons. Identifying the best possible approach for HA could lead to shorter hospital admission, faster rehabilitation, better functional outcomes, lower morbidity and mortality and improvement in patient independence. Consequently healthcare costs related to a hip fracture could be reduced.

As of today the clinical results, reoperation rate and the morbidity have improved significantly in hemiarthroplasty treatment for dislocated femoral neck fractures. However, patients are primarily operated with the lateral approach, although inferior results are reported compared to posterior and anterior approaches. RCT´s from Ugland et al and Mjaaland have shown increased incidence of limping, lateral thigh pain and inferior PROM´s in patients operated with the direct lateral approach compared to patients operated with anterior approaches.

A meta-analysis regarding hemiarthroplasty and surgical approaches from 2018 concluded that high-quality comparative studies are needed to further substantiate the preferred anatomic route for hemiarthroplasty in older femoral neck fracture patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 70 and 90 years of age
* Displaced FNF
* Ability to walk with or without a walking aid prior to falling
* Patients having Sorlandet Hospital as primary service provider for orthopaedic trauma
* Provision of informed consent by patient or proxy
* Low energy fracture (fall from standing height, no other major trauma)

Exclusion Criteria:

* Dementia
* Fractures in pathologic bone
* Patients not suited for HA (i.e., inflammatory arthritis, severe osteoarthritis)
* Associated major injuries of the lower extremity ( i.e., ipsilateral or contralateral fractures of the foot, ankle, tibia, fibula or femur)
* Retained hardware around the affected hip that will interfere with arthroplasty
* Sepsis or local infection

Ages: 70 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2022-01-21 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score | 2 years
  The posterior SPAIRE and the anterior approach in HA for femoral neck fractures results in equivalent patient reported outcome measured by Harris Hip Score.

SECONDARY OUTCOMES:
Bone Mineral Density | 2 years
  The posterior SPAIRE and the anterior approach in HA for femoral neck fractures results in equivalent postoperative changes in bone mineral density measured by dual-energy X-ray absorptiometry (DXA).
Muscle damage | 2 years
  The posterior SPAIRE and the anterior approach in HA for femoral neck fractures results in equivalent postoperative changes in biochemical muscle damage measured by Creatin Kinase (CK)
Muscle damage | 2 years
  The posterior SPAIRE and the anterior approach in HA for femoral neck fractures results in equivalent postoperative changes in clinical muscle damage measured by TUG-test
Muscle damage | 2 years
  The posterior SPAIRE and the anterior approach in HA for femoral neck fractures results in equivalent postoperative changes in clinical muscle damage measured by Trendelenburg test
Muscle damage | 2 years
  The posterior SPAIRE and the anterior approach in HA for femoral neck fractures results in equivalent postoperative changes in clinical muscle damage measured by muscle strength
Health-related quality of life (HRQoL) | 2 years
  The posterior SPAIRE and the anterior approach in HA for femoral neck fractures results in equivalent health-related quality of life (HRQoL) measured by HOOS
Health-related quality of life (HRQoL) | 2 years
  The posterior SPAIRE and the anterior approach in HA for femoral neck fractures results in equivalent health-related quality of life (HRQoL) measured by Eq-5d
Health-related quality of life (HRQoL) | 2 years
  The posterior SPAIRE and the anterior approach in HA for femoral neck fractures results in equivalent health-related quality of life (HRQoL) measured by Visual Analog Score (VAS)
Radiographic stem positioning | 2 years
  The posterior SPAIRE and the anterior approach in HA for femoral neck fractures results in equivalent radiographic stem positioning.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nordsletten, MD,PhD,Professor, Study Director — Oslo University Hospital
Locations (2):
- Norway (2):
  - Sorlandet Hospital, Arendal
  - Sorlandet hospital, Kristiansand